CLINICAL TRIAL: NCT01390571
Title: A Cancer Research UK Phase I Trial of Olaparib (AZD2281), an Oral PARP Inhibitor, in Combination With Extended Low-Dose Oral Temozolomide in Patients With Relapsed Glioblastoma
Brief Title: Olaparib and Temozolomide in Treating Patients With Relapsed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000702605; CRUK-CR0901-11; EUDRACT-2010-018615-15
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — olaparib; Temozolomide; Gene Expression Profiling

INTERVENTIONS:
Drug: olaparib
Drug: temozolomide
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: diffusion-weighted magnetic resonance imaging
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Olaparib may help temozolomide kill more tumor cells by making tumor cells more sensitive to the drug.

PURPOSE: This phase I trial is studying the side effects and best dose of olaparib and temozolomide in treating patients with relapsed glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether olaparib crosses the blood-brain barrier (BBB) and achieves tumor penetration in patients with relapsed glioblastoma. (Stage 1)
* To determine the safety and tolerability of the combination of olaparib and temozolomide in patients with relapsed glioblastoma. (Stage 2)

Secondary

* To assess BBB disruption and BBB permeability in patients with relapsed glioblastoma. (Stage 1 and stage 2 maximum-tolerated dose [MTD] expansion cohort)
* To assess the possible anti-tumor activity of the combination of olaparib and temozolomide in patients with relapsed glioblastoma. (Stage 2)

Tertiary

* To assess biological markers as possible predictors of olaparib efficacy in patients with glioblastoma.
* To optimize techniques for measuring DNA damage responses to PARP inhibition in tumor tissue.
* To determine plasma concentration of olaparib at the time of surgery in patients with glioblastoma.
* To evaluate the PARP inhibition at the time of surgery in peripheral blood mononuclear cells (PBMCs).

OUTLINE: This is a multicenter, dose-escalation study.

* Stage 1: Patients receive fixed-dose oral olaparib twice daily for 3 days prior to resection and then receive a dose of oral olaparib on the morning of the resection. After the surgical resection, patient receive standard of care treatment. Patients undergo dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) and diffusion-weighted imaging (DWI) scans to assess the disruption and permeability of the blood-brain barrier (BBB).

Stage 1 is complete and it was proven that olaparib can cross the BBB and achieve tumour penetration in glioblastoma patients.

* Stage 2: Patients receive escalating doses of oral olaparib once or twice daily for 3 days prior to resection and then receive a dose of oral olaparib on the morning of the resection. After recovery from surgery, patients receive oral olaparib once or twice daily and oral temozolomide once daily on days 1-42. Treatment repeats every 8 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients may receive 3 additional courses of treatment in the absence of disease progression.

Once the maximum tolerated dose (MTD) is established, 10 more patients are treated at the MTD as stage 2 MTD expansion cohort. These patients also undergo DCE-MRI and DWI scans.

All patients undergo blood collection periodically for pharmacokinetic and pharmacodynamic studies.

After completion of study treatment, patients are followed up for 28 days and then monthly until resolution of study drug-related adverse events.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade IV glioblastoma
* Radiological diagnosis of recurrent or progressive disease according to Response Assessment in Neuro-Oncology Working Group (RANO) criteria, which is suitable for palliative resection
* Must have an adequate amount of tumor tissue available
* Previously received first-line treatment with radical radiotherapy, or chemoradiation followed by adjuvant chemotherapy

  * No prior chemotherapy for recurrent disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 12 weeks
* Hemoglobin ≥ 10.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT or AST ≤ 2.5 times ULN
* Calculated creatinine clearance ≥ 50 mL/min OR isotope clearance measurement ≥ 50 mL/min (uncorrected)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use one (male) or two (female) highly effective forms of contraception 4 weeks prior to, during, and for 6 months after completion of study therapy
* Able to swallow and retain oral medications
* Not at high medical risk due to non-malignant systemic disease, including active uncontrolled infection
* No known hepatitis B, hepatitis C, or HIV seropositivity
* No concurrent congestive heart failure, prior history of NYHA class III-IV cardiac disease, prior history of cardiac ischemia, or prior history of cardiac arrhythmia within the past 12 months
* No grand mal seizures occurring ≥ 3 times per week over the past month
* No gastrointestinal disorders likely to interfere with absorption of the study medication
* No known hypersensitivity to any of the components of olaparib
* No known hypersensitivity to temozolomide (TMZ) or any of its components, or to dacarbazine (DTIC) (for patients enrolled in stage 2 study only)
* No known lactose intolerance (for patients enrolled in the stage 2 study only)
* No metal fragments in the eyes (shrapnel or bullet injuries are excluded on the basis of their unsuitability to undergo MRI scans)
* No other condition which, in the Investigator's opinion, would not make the patient a good candidate for the clinical trial

EXCLUSION CRITERIA:

* See Disease Characteristics
* No ongoing toxic manifestations from previous treatments except for alopecia or grade 1 toxicities which, in the opinion of the Investigator and the Drug Development Office (DDO), should not exclude the patient
* At least 12 weeks since prior radiotherapy, endocrine therapy, or immunotherapy
* At least 6 weeks since prior major surgery
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior immunizations with live vaccines (or expected to receive vaccines during the trial and up to at least 6 months after receiving last study treatment), including BCG and yellow fever vaccines
* No prior PARP inhibitors, including olaparib
* No prior major thoracic or abdominal surgery from which the patient has not yet recovered
* No prior heart surgery
* No pacemakers
* No change to systemic steroids dose within 5 days prior to enrollment (i.e., must be on a stable dose at time of enrollment and remain on a stable dose throughout the treatment period)
* No herbal supplements and/or ingestion of foods known to modulate CYP3A4 enzyme activity from time entered on screening period until 28 days after the last dose of study medication
* No concurrent drugs known to be potent inducers of CYP3A4, including phenytoin, carbamazepine, phenobarbital, rifampicin, rifapentine, rifabutin, nevirapine, modafinil, or St. John wort (wash-out period for phenobarbital is 5 weeks, 3 weeks for all others)
* No concurrent drugs known to be potent inhibitors of CYP3A4, including ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin, or nelfinavir (wash-out period is 1 week)
* No concurrent or planned participation in another interventional clinical study

  * Participation in an observational study is acceptable
* No concurrent warfarin (patients requiring anticoagulation should be given subcutaneous low molecular weight heparin)
* No other concurrent anticancer therapy (including radiotherapy) or investigational drugs

  * No blood transfusions within 4 weeks prior to study start of features suggestive of myelodysplasia or AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-07; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Detection of olaparib in tumor tissue using liquid chromatography mass spectrometry (LC-MS) seen in at least 1 out of the 6 patients treated in stage 1 of the study
Maximum-tolerated dose of olaparib in combination with temozolomide (stage 2)
Toxicity profile and dose-limiting toxicity as assessed by NCI CTCAE Version 4.02 (stage 2)

SECONDARY OUTCOMES:
Measurement of blood-brain barrier (BBB) disruption and permeability biomarkers by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) and diffusion-weighted imaging (DWI) (stage 1 and stage 2 MTD expansion cohort)
Progression-free survival at 6 months post-surgery as assessed by the Response Assessment in Neuro-Oncology Working Group (RANO) criteria from conventional MRI and clinical assessment (stage 2)

OTHER OUTCOMES:
Gene copy number analysis of DNA repair genes
Quantification of DNA repair gene expression
Measurement of methylation of the MGMT promoter gene by bisulfite modification of DNA and pyrosequencing
Measurement of microsatellite instability by Multiplex PCR
Measurement of mismatch repair (MMR) gene expression by quantitative real time polymerase chain reaction (QRT-PCR) analysis
Measurement of phosphatase and tensin homolog (PTEN) protein and gene expression
Quantification of global DNA strand breaks in tumour tissue by Immunostaining for γH2AX
Measurement of Rad51 foci and nuclear staining intensity as markers of homologous recombination (HR) repair activity
Plasma levels of olaparib measured by LC-MS
PARP inhibition measured by validated assays
Detection of olaparib in tumour margin tissue using LC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Chalmers, Prof, Principal Investigator — Beatson West of Scotland Cancer Centre
Locations (7):
- United Kingdom (7):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Christie Hospital, Manchester, England
  - Royal Marsden Hospital, Sutton, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Queen Elizabeth Hospital, Birmingham
  - Western General Hospital, Edinburgh